CLINICAL TRIAL: NCT04390932
Title: The Impact of Therapeutic Alliance on Clinical Outcomes in Patients With Symptomatic Knee Osteoarthritis. A Randomized Clinical Trial Protocol.
Brief Title: The Impact of Therapeutic Alliance in the Rehabilitation of Knee Osteoarthritis.
Acronym: ALLIANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Catolica de Temuco (Other)
Responsible Party: Principal Investigator, Iván Alejandro Cuyul Vásquez, Associate Professor, Universidad Catolica de Temuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCTKINE2020
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: Therapeutic Alliance; Professional-Patient Relations; Pain; Osteoarthritis; Exercise Therapy.
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Opaque sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced TA (Experimental): Therapeutic exercise protocol accompanied by an enhanced TA.
  Interventions: Other: Enhanced TA; Other: Therapeutic exercise protocol.
- Neutral therapeutic alliance (Active Comparator): Therapeutic exercise protocol accompanied by an limited TA
  Interventions: Other: Limited TA; Other: Therapeutic exercise protocol.

INTERVENTIONS:
Other: Enhanced TA — The enhanced TA is characterized by the personalization of the conversation, the verbalization of a joint participation in the process, the full presence of the therapist in the development of the exercise protocol, and the inclusion of behaviors such as active listening, empathy, and encouragement. In addition, therapist's body language transmits confidence, security, and attention.
  Arms: Enhanced TA
Other: Limited TA — The limited TA does not consider the personalization of the conversation, uses a unidirectional verbalization and is imperative about the instructions provided to the participant, the therapist is intermittently absent during the therapeutic exercise sessions and uses a neutral or negative nonverbal language cues.
  Arms: Neutral therapeutic alliance
Other: Therapeutic exercise protocol. — Three 45-60 minute sessions of supervised therapeutic exercise (combination of aerobic, isometric, and isotonic exercise) delivered within a one-week period.

SUMMARY:
The therapeutic alliance (TA) is the working relationship or positive social bond between the patient and the therapist. TA is based on collaboration, communication, empathy of the therapist and mutual respect. Fostering an enhanced therapeutic alliance is a low-cost, therapist-dependent strategy that can accompany any clinical intervention. Growing evidence suggests that the TA plays a pivotal role in clinical outcomes in psychotherapy, medicine and physiotherapy interventions for chronic low back pain. On the other hand, therapeutic exercise is an economic, accessible and simple intervention strategy that has proven to be effective and safe to decrease pain and improve physical function in people with knee osteoarthritis (OA). To date, the role of TA in the management of knee OA is unknown. We hypothesized that a therapeutic exercise protocol accompanied by an enhanced TA could reduce the severity of symptoms and improve function in patients with symptomatic knee OA.

DETAILED DESCRIPTION:
The objective of this randomized clinical trial will be to determine the effects of different levels of TA during the application of a therapeutic exercise program on pain intensity, pressure pain thresholds and function in patients with symptomatic knee OA.

ELIGIBILITY:
Inclusion Criteria:

- People aged 45 to 65 years with a clinical and radiographic diagnosis of knee osteoarthritis (grade I-III according to Kellgren and Lawrance), symptomatic with pain intensity between 3 and 8 points in the PI-NRS with at least 3 months duration, resulting in a mild to moderate level of disability (WOMAC).

Exclusion Criteria:

- People with other musculoskeletal, neurological, or immune conditions that cause pain or functional limitation in the lower extremities (hip osteoarthritis, patellar tendinopathy, sprains, radiculopathies, rheumatoid arthritis, systemic lupus erythematosus), history of trauma less than a year ago ( knee fractures, meniscal or ligament tears) or surgery of any kind on the lower extremity. Knee mobility less than 90º flexion. People in treatment with oral or intra-articular corticosteroids, antibiotics or exogenous opioids of any kind, with unstable cardiovascular, respiratory, systemic or metabolic conditions that do not allow physical exercise.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 48 hours post intervention
  Change in numerical pain rating scale (PI-NRS)
Pressure pain thresholds | 48 hours post intervention
  Change in pressure algometry

OTHER OUTCOMES:
Lower limb function | Only in the evaluation of the baseline.
  WOMAC physical function section
Therapeutic alliance | 48 hours post intervention
  Work Alliance Sub-scale of the Rehabilitation Expectations Scale (PRES)
Expectations level | Only in the evaluation of the baseline.
  Credibility and Expectations Questionnaire
Conditioned pain modulation | Only in the evaluation of the baseline.
  Change in pressure algometry after application of cold inmmersion test
Anxiety and depression | Only in the evaluation of the baseline.
  Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Iván A Cuyul-Vásquez, Principal Investigator — Universidad Catolica de Temuco
Locations (1):
- UC Temuco, Temuco, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuyul-Vasquez I, Fuentes C J. Effects of therapeutic alliance on clinical outcomes in patients with symptomatic knee osteoarthritis undergoing an exercise program: A randomized clinical trial protocol. Medwave. 2021 Apr 16;21(3):e8160. doi: 10.5867/medwave.2021.03.8159. PMID 33956775